CLINICAL TRIAL: NCT05598853
Title: Intrathecal Administration of Anti-PD1/Anti-CTLA-4 in Combination With Systemic Combination of Anti-PD1/Anti-CTLA-4 in Patients With NSCLC Without Oncogenic Driver Mutation or Melanoma and Newly Diagnosed Leptomeningeal Metastasis: a Multicentric Phase I Study
Brief Title: Intrathecal Double Checkpoint Inhibition
Acronym: IT-IO
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IT-IO (CA209-6K7)
Record Dates: First submitted 2022-10-11; First posted 2022-10-28 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Leptomeningeal Metastasis; Non-small Cell Lung Cancer Stage IV; Melanoma Stage IV
Keywords: intrathecal; immunotherapy
MeSH Terms: conditions — Meningeal Carcinomatosis; Carcinoma, Non-Small-Cell Lung; Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Intrathecal nivolumab and intrathecal ipilimumab (Experimental): The experimental treatment will be combined from cycle 2 with systemic nivolumab and systemic ipilimumab
  Interventions: Drug: intrathecal nivolumab and intrathecal ipilimumab

INTERVENTIONS:
Drug: intrathecal nivolumab and intrathecal ipilimumab — Patients shall be treated with a fixed dose of intrathecal nivolumab and increasing doses of intrathecal ipilimumab. From cycle 2, patients will receive systemic nivolumab/ipilimumab in addition to intrathecal treatment. Systemic nivolumab/ipilimumab corresponds to the current standard of care for non-small cell lung cancer and for melanoma patients.

SUMMARY:
The objective of the present study is to determine the feasibility and to explore anti-tumor activity of intrathecal double immune checkpoint inhibition for patients with newly diagnosed leptomeningeal metastases from non-small cell lung cancer without driver mutation or melanoma.

DETAILED DESCRIPTION:
The treatment regimen within the IT-IO study consists of intrathecal administration of nivolumab/ipilimumab in combination with systemic combined nivolumab/ipilimumab.

The scheme of administration of systemic nivolumab/ipilimumab corresponds to the current standard of care for non-small cell lung cancer and for melanoma patients.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed confirmed or probable leptomeningeal metastases according to European Association of Neuro-Oncology (EANO) - European Society for Medical oncology (ESMO) criteria (Le Rhun et al., 2017).
* Histologically confirmed (from primary tumor or from a metastatic lesion, including in the brain) non-small cell lung cancer without actionable oncogenic driver mutation or melanoma. Programmed death-ligand 1 (PD-L1) expression status (from primary tumor or from a metastatic lesion, including brain) is optional, but should be documented if available

  * Requirements for patients with non-small cell lung cancer: non-small cell lung cancer without a specified targetable oncogenic driver alteration: sensitising Epidermal Growth Factor Receptor (EGFR) mutation (exon 19-del and 21-L858R), anaplastic lymphoma kinase (ALK) or ROS proto-oncogene-1 (ROS1) rearrangement.
* Clinically eligible for systemic immunotherapy with nivolumab and ipilimumab at the time of enrolment as judged by the investigator. If already initiated, the systemic treatment must be well tolerated, without common terminology criteria for adverse events (CTCAE) grade 3 or more toxicity, and there must be no evidence of systemic progression and no indication for whole brain radiotherapy. Intrathecal immunotherapy alone may be acceptable for exceptional patients after discussion with the coordinators of the study. Systemic immunotherapy can be started later in these patients based on investigator decision.
* Patients previously treated with systemic chemotherapy must have received the last dose at least 21 days prior to treatment initiation, patients who have received another investigational agent must have received the last treatment at least 14 days prior to treatment initiation.
* Age of 18 years or older on day of signing informed consent, female or male.
* Karnofsky performance status of 60 or more.
* Life expectancy >8 weeks. Patients with rapidly progressive systemic disease are not eligible.
* Patients may receive steroids to control symptoms related to central nervous system involvement, but the dose must be stable or decreasing and < 4 mg per 24 hours of dexamethasone (or equivalent) in the last 7 days. Patients should experience stability of neurological symptoms for at least 7 days. Physiologic replacement doses of steroids are permitted.
* Cerebrospinal MRI criteria (on the baseline MRI, performed within 14 days prior to study treatment initiation)

  * MRI can be normal or can show leptomeningeal metastases, including nodules <0.5 cm diameter largest diameter (or more if stereotactic radiosurgery is planned)
  * No evidence of cerebrospinal fluid flow obstruction at the discretion of the investigator
  * Co-existing asymptomatic brain metastases <2 cm diameter are permitted. Larger asymptomatic or oligosymptomatic brain metastases are permitted if they are planned to be treated by stereotactic radiosurgery
* Central nervous system radiotherapy criteria:

  * Focal brain radiotherapy by stereotactic radiotherapy is allowed for meningeal nodules > 5 mm diameter or concomitant brain metastases. The treated lesions cannot be used as a target for the evaluation of the study treatment
  * Prior brain focal radiotherapy for central nervous system metastases is permitted if completed at least 14 days prior to enrolment, but the treated lesions cannot be used as a target for the evaluation of the study treatment
  * Planned whole brain radiotherapy is not allowed
  * Prior whole brain radiotherapy for brain metastases is permitted if terminated at least 3 months prior enrolment.
  * Planned or prior craniospinal irradiation is not allowed
* Women of childbearing potential, including women who had their last menstruation in the last 2 years, must have a negative urinary or serum pregnancy test within 24 hours before the first dose of study treatment.
* Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and return for the required assessments.
* Written informed consent for study participation must be signed and dated by the patient and the investigator prior to any study-related intervention.

Exclusion Criteria:

* Leptomeningeal metastases related to primary tumors other than non-small cell lung cancer without driver mutation or melanoma.
* Inability to undergo craniospinal MRI evaluation.
* Progressive parenchymal brain metastases thought to require whole brain radiotherapy.
* Contra-indication to lumbar puncture or to implantation of a ventricular device.
* Prior intrathecal chemotherapy, intrathecal immunotherapy or intrathecal targeted therapy.
* Ventriculo-peritoneal shunt (except if intrathecal therapy is administered via a ventricular device with an ON/OFF option).
* Condition requiring systemic treatment with either corticosteroids (> 4 mg daily dexamethasone equivalents) or other immunosuppressive medications within 7 days of study drug administration. Inhaled or topical steroids and adrenal replacement doses < 10 mg daily prednisone equivalents are permitted in the absence of active autoimmune disease.
* Patients with a history of pneumonitis or previous non-hematological grade >2 toxicity under previous immunotherapy treatment.
* Active infection (systemic or central nervous system) within 7 days prior to initiation of the study drug.
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Known positive test for hepatitis B virus surface antigen (HBV sAg) or hepatitis C virus ribonucleic acid (HCV antibody) indicating acute or active chronic infection.
* Known history of testing positive for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) even if fully immunocompetent on antiretroviral therapy due to the unknown effects of HIV on the immune response to combined nivolumab plus ipilimumab or the unique toxicity spectrum of these drugs in patients with HIV infection.
* Use of vaccines containing live virus for prevention of infectious disease within 12 weeks prior to study drug.
* History of allergy to study drug components and history of severe hypersensitivity reaction to any monoclonal antibody.
* Concurrent treatment with other systemic cancer-derived pharmacotherapies is not allowed. No other concomitant intrathecal therapy is allowed.
* Any investigational anticancer therapy other than those under investigation in this study.
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
* Intention to become pregnant during the course of the study. Women who are pregnant.
* Women who are breast feeding and who do not agree to discontinue nursing prior to the first study treatment and for the period defined in the protocol.
* Sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method during the study.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Estimated)
Dates: Start 2022-11-25 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Recommended phase II dose of intrathecal (IT) nivolumab/ipilimumab followed by IT nivolumab/ipilimumab plus systemic nivolumab/ipilimumab | 3 weeks
  Determination of the maximum tolerated dose or the recommended phase II dose for combined intrathecal immunotherapy

SECONDARY OUTCOMES:
steroid intake | through study completion, an average of 1 year
  steroid intake in mg dexamethasone at each assessment
compartmental efficacy (PFS) of nivolumab/ipilimumab combined with systemic nivolumab/ipilimumab | through study completion, an average of 1 year
  progression free survival in months by compartments level (leptomeningeal compartment, brain compartment, central nervous system compartment, extra-central nervous system compartment, overall compartment)
compartmental efficacy (response) of nivolumab/ipilimumab combined with systemic nivolumab/ipilimumab | through study completion, an average of 1 year
  response rate in percentage by compartments level (leptomeningeal compartment, brain compartment, central nervous system compartment, extra-central nervous system compartment, overall compartment)
efficacy of nivolumab/ipilimumab combined with systemic nivolumab/ipilimumab | through study completion, an average of 1 year
  overall survival in months
prognostic factors | through study completion, an average of 1 year
  association between survival and prognostic factors. The list of items to analyze will be determined prior to the analysis to consider potential new data available in the literature. The analysis will be performed in the whole population, per cerebrospinal fluid cytology assessment at diagnosis (positive cerebrospinal fluid cytology versus equivocal or negative cerebrospinal fluid cytology); per tumor entity (non-small cell lung cancer versus melanoma)

CONTACTS AND LOCATIONS:
Locations (3):
- Switzerland (3):
  - University Hospital Zurich, Zurich, Canton of Zurich
  - University Hospital Basel, Basel
  - University Hospital Geneva, Geneva

IPD SHARING:
Plan to Share IPD: No